CLINICAL TRIAL: NCT06180122
Title: The Use and Reproducibility of Duplex Ultrasound to Provide Indices of Left Common Iliac Vein (CIV) Diameter, to Aid and Improve the Diagnosis of May Thurner Syndrome (MTS) in Patients Presenting With Unexplained Left Leg Swelling
Brief Title: The Use and Reproducibility of Duplex Ultrasound to Provide Indices of Left Common Iliac Vein Diameter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23CX8043
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: May-Thurner Syndrome
MeSH Terms: conditions — May-Thurner Syndrome | interventions — Ultrasonography, Doppler, Duplex

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptomatic Group (Other): Participants who are suffer from unexplained left leg swelling.
  Interventions: Diagnostic Test: Duplex ultrasound
- Asymptomatic Group (Other): Participants who do not suffer from unexplained left leg swelling
  Interventions: Diagnostic Test: Duplex ultrasound

INTERVENTIONS:
Diagnostic Test: Duplex ultrasound — Vascular ultrasound scan of the left common iliac vein

SUMMARY:
The goal of this feasibility/pilot study is to investigate whether or not vascular ultrasound can be used to aid the diagnosis of May Thurner Syndrome, in adult patients presenting to the vascular department with unexplained left leg swelling. The main research objective it aims to answer are:

* The diameter variation of the left common iliac vein based on posture, using duplex ultrasound.
* To determine inter- and intra-observer variation of the diameter measurement of the left common iliac vein using duplex ultrasound.

Participants will have an ultrasound scan performed on their abdomen by three different clinical vascular scientists, and will have each scan performed whilst lying supine on an examination couch and again when the couch is tilted to 45 degrees.

Researchers will compare the results of symptomatic patients to asymptomatic patients, to see if there is a difference in the diameter of the left common iliac vein between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* Participant has the capacity to consent
* Participant is required to have a vascular ultrasound scan in the vascular ultrasound department
* Participant is 18 years of age or older at the start of the study.

Exclusion Criteria:

* Previous iliac vein intervention or treatment for iliac vein disease
* Previous diagnosis of iliac vein thrombus
* Pregnancy
* Unable to provide appropriate informed consent
* The participant does not require a vascular ultrasound as part of their routine care
* Under 18 years of age at the start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from Vascular Outpatients clinic at Charing Cross Hospital between March 2024 and May 2024.
Pre-assignment Details: Questionnaire used to obtain a medical history taken from patient on morning of ultrasound scan, to determine which study group the participant should be allocated to (symptomatic or asymptomatic).
Groups:
- Symptomatic Group: Participants who suffer from unexplained left leg swelling.
Period: Overall Study
Arm/Group | Symptomatic Group | Asymptomatic Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symptomatic Group | Asymptomatic Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Full Range); unit: Years] — Age of each participant recorded, mean age of the each group provided
  Years | 52 [25 to 78] | 56 [29 to 78] | 54 [25 to 78]
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants of each sex provided
  Participants
    Female | 13 | 9 | 22
    Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Participants asked to describe their ethnicity, a range of results provided
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 20 | 20 | 40
    Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Full Range); unit: kg/m^2] — Height and weight taken from each participant, BMI calculated
  kg/m^2 | 29 [19 to 47] | 25 [15 to 36] | 27 [15 to 47]

OUTCOME MEASURES:

1. Primary Outcome: Left Common Iliac Vein Diameter
Description: The diameter measurement (in mm) of the left common iliac vein in adults referred to the vascular ultrasound department.
Time Frame: Baseline
Population: Data could not be obtained from one participant in the symptomatic group due to non-visualization of the common iliac vein
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | Symptomatic Group | Asymptomatic Group
Number analyzed (Participants) | 19 | 20
Millimeters (mm) | 7.5 (2.9) | 7.7 (2.3)

2. Secondary Outcome: Inter-and Intra-operator Variation of the Diameter Measurement of the Left Common Iliac Vein
Description: The inter- and intra-operator variation of the diameter measurement of the left common iliac vein using duplex ultrasound, in adults referred to the vascular ultrasound department. Three different scientists took three measurements each of the common iliac vein. The results from the three scientists were compared to determine inter-operator variation, and the results from one scientist each were compared to determine intra-operator variation.
Time Frame: Baseline
Measure: Number (95% Confidence Interval); unit: ICC - Reliability/descriptive statistic
Groups:
- Interoperator Variability: Comparison of variability of measurements taken by each operator
- Intraoperator Variability: Comparison of variability of measurements taken between each of the three operators
Arm/Group | Interoperator Variability | Intraoperator Variability
Number analyzed (Participants) | 39 | 39
ICC - Reliability/descriptive statistic | 0.67 [0.60 to 0.72] | 0.92 [0.90 to 0.93]

ADVERSE EVENTS:
Time Frame: On the study day / day of the ultrasound scan
Description: No difference
Arm/Group | Symptomatic Group | Asymptomatic Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Limitation due to non-visualization of the CIV in some participants - In one participant no readings/data could be obtained, and in three participants only partial data could be obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT06180122/Prot_SAP_000.pdf